CLINICAL TRIAL: NCT06307704
Title: Intraoperative Bedside Lung-ultrasound Use to Optimize Positive End-expiratory Pressure for Elective Robotic-assisted Radical Prostatectomy or Cystectomy Patients: a Randomized Controlled Trial
Brief Title: Lung US for PEEP Optimization in Robotic Radical Prostatectomy or Cystectomy Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nazmy Edward Seif (Other)
Responsible Party: Sponsor-Investigator, Nazmy Edward Seif, Clinical Professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: LUSPEEPORRPC
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer; Urinary Bladder Cancer; Surgery; Positive End Expiratory Pressure; Lung Ultrasound
Keywords: Radical Cystectomy; Radical Prostatectomy; Robotic; Anesthesia; Lung-Ultrasound; Positive End Expiratory Pressure
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US - PEEP group (Experimental): Lung Ultrasound - guided Positive End Expiratory Pressure group
  Interventions: Procedure: Lung Ultrasound - guided Stepwise PEEP; Procedure: Standard Ventilation Protocol
- Standard group (Active Comparator): Standard Ventilation group
  Interventions: Procedure: Standard Ventilation Protocol

INTERVENTIONS:
Procedure: Lung Ultrasound - guided Stepwise PEEP — After endo-tracheal intubation; A PEEP of 4 cmH2O will be initially used till 5 min after pneumoperitoneum. Then The PEEP will be adjusted in a stepwise approach after performing bedside lung ultrasound. The PEEP will be increased by 2 cmH2O until no lung collapse is detected. Lung ultrasound will be repeated 5 min after every change in the PEEP with a maximal PEEP of 12 cmH2O.
  Arms: US - PEEP group
Procedure: Standard Ventilation Protocol — Volume-controlled ventilation (VCV) mode; with a tidal volume of 6 mL/kg of ideal weight, inspiratory : expiratory ratio 1: 2, PEEP 4 cmH2O, respiratory rate adjusted to keep end-tidal carbon dioxide tension (EtCO2) between 35 and 40 mm Hg, and inspired oxygen fraction of 50%.

SUMMARY:
There is an increasing trend in the use of robotic-assisted radical prostatectomy or cystectomy (RARPC).

Preventing lung atelectasis without inducing overdistention of the lung is challenging. Many studies tried to optimize PEEP titration by using methods such as dead space fraction guided and static pulmonary compliance directed techniques, or by using electrical impedance tomography. However, the use of these methods is limited by inaccuracy and the need for sophisticated devices.

Bedside Lung ultrasound is fast, easy and economic technique that is gaining interest in the operating room. Ultrasound-guided PEEP titration has been used in bariatric surgeries (different position and usually shorter procedure time) and proved effective in improving oxygenation, compliance and reducing the incidence of postoperative pulmonary atelectasis and hypoxia without causing hemodynamic instability.

The aim of this study is to evaluate the effectiveness of intraoperative individualized lung ultrasound-guided stepwise PEEP optimization in patients undergoing RARPC on oxygenation, intraoperative and early postoperative pulmonary complications.

ELIGIBILITY:
Inclusion Criteria:

* ASA I, II & III.
* Normal respiratory functions or mild lung disease.

Exclusion Criteria:

* BMI more than 40.
* Moderate to severe obstructive pulmonary disease (FEV1 < 80% of predicted).
* Moderate to severe restrictive pulmonary disease (TLC < 70% of predicted).
* Severe pulmonary hypertension (mean PAP>55).
* Previous lung surgery.
* Decompensated cardiac disease (NYHA 3 or 4).
* Patients who received invasive mechanical ventilation within the last 30 days before surgery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Post-operative lung consolidation | 24 hours
  Presence (or not) of post-operative lung consolidation detected by lung ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Ashgan R Ali, MD, Study Chair — Kasr Al-Ainy Hospital, Faculty of Medicine, Cairo University; Nazmy S Mikhael, MD, Principal Investigator — Kasr Al-Ainy Hospital, Faculty of Medicine, Cairo University; Mustafa E Mohamed, MD, Study Director — Kasr Al-Ainy Hospital, Faculty of Medicine, Cairo University
Locations (1):
- Cairo University Hospitals, Cairo, Egypt